CLINICAL TRIAL: NCT00566020
Title: Study SCA106052, a Clinical Evaluation of BW430C (Lamotrigine) in Bipolar I Disorder- Long-term Extension Study (Extension of Study SCA104779 (NCT00550407))
Brief Title: A Clinical Evaluation Of BW430C (Lamotrigine) In Bipolar I Disorder- Long-term Extension Of Study SCA104779 (NCT00550407) -
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SCA106052
Record Dates: First submitted 2007-11-28; First posted 2007-11-30 (Estimated); Results first posted 2011-07-27 (Estimated); Last update posted 2017-04-04 (Actual); Status verified 2017-03

CONDITIONS: Bipolar Disorder
Keywords: Open-label extension; Tolerability; Lamotrigine; Safety; Bipolar I disorder
MeSH Terms: conditions — Bipolar Disorder | interventions — Lamotrigine

ARMS (1):
- Lamotrigine (Experimental): study drug
  Interventions: Drug: BW430C (lamotrigine)

INTERVENTIONS:
Drug: BW430C (lamotrigine) — lamotrigine 50mg/day-400mg/day

SUMMARY:
This study is planned to assess the long-term safety of lamotrigine in Japanese patients with bipolar I disorder who will continue into the 52-week extension upon completion of a double-blind comparative study (Study No.: SCA104779 (NCT00550407)), i.e. the patients who receive the addition of any additional treatment to intervene in a mood episode in the double-blind phase or the patients completing the double-blind phase.

ELIGIBILITY:
Inclusion Criteria:

* Of subjects participating in the preceding double-blind study, those who are judged by the investigator/sub-investigator to have well tolerated the double-blind treatment and to be eligible for the 52-week extension treatment
* Sex: either sex. Female of child-bearing potential will be eligible for inclusion in this study. However they have to have a negative pregnancy test at the start of this study, agree to further pregnancy testing at the time points determined in study assessments and procedures and practice one of the following methods of contraception from the start of this study until the end of the follow-up examination:

Abstinence

Oral contraceptive, either combined or progestogen alone (except during the Dosage Adjustment Phase)

Injectable progestogen

Implants of levonorgestrel

Estrogenic vaginal ring (except during the Dosage Adjustment Phase)

Percutaneous contraceptive patches (except during the Dosage Adjustment Phase)

Intrauterine device (IUD) or intrauterine system (IUS) that meets the SOP effectiveness criteria as stated in the product label

Male partner sterilization (vasectomy with documentation of azoospermia) prior to the female subject's entry into the study, and this male is the sole partner for that subject

Double barrier method: condom or occlusive cap (diaphragm or cervical / vault caps) plus spermicidal agent (foam / gel / film / cream / suppository)

* In/Out patient: Either
* Informed consent: the subject capable of giving written informed consent

Exclusion Criteria:

* Has a score of 3 or more on item of the HAM-D related to suicide or is at a high suicidal risk in the judgment of the investigator/sub-investigator
* Has a history of severe rash or rash due to anti-epileptic drugs
* Patients with severe hepatic/renal/cardiac/pulmonary disorder or hematopoietic disorder. The severity refers to Grade 3 according to "the Classification of the Severity of Adverse Experiences" (PAB/SD Notification No. 80, dated 29 June 1992)
* Patients have less than 5 years of remission history from clinically significant malignancy (other than e.g. basal cell or squamous cell skin cancer, in-situ carcinoma of cervix or prostate CA in situ)
* Patients with chronic hepatitis typeB and /or typeC which is positive of hepatitis B surface antigen （HBsAg）and/or hepatitis C antibody
* Has an acute or chronic illness likely to impair drug absorption, distribution, metabolism or excretion or has any unstable physical symptoms likely to require hospitalisation during participation in the study
* Female patients who are pregnant or lactating, who may be pregnant, or who plan for pregnancy during the study
* Has a history or current diagnosis of epilepsy
* Has received an investigational drug within 30 days of screening
* Patients with a history of drug allergy to any ingredient of the test-drug
* Patients whom the investigator or sub-investigator considers ineligible for the study

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 92 (Actual)
Dates: Start 2008-05; Primary Completion 2010-10 (Actual); Study Completion 2010-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (20):
- Japan (20):
  - GSK Investigational Site, Aichi
  - GSK Investigational Site, Chiba
  - GSK Investigational Site, Fukuoka
  - GSK Investigational Site, Gunma
  - GSK Investigational Site, Hiroshima
  - GSK Investigational Site, Hokkaido
  - GSK Investigational Site, Ibaraki
  - GSK Investigational Site, Kanagawa
  - GSK Investigational Site, Kumamoto
  - GSK Investigational Site, Kyoto
  - GSK Investigational Site, Mie
  - GSK Investigational Site, Nara
  - GSK Investigational Site, Okayama
  - GSK Investigational Site, Osaka
  - GSK Investigational Site, Ōita
  - GSK Investigational Site, Saga
  - GSK Investigational Site, Saitama
  - GSK Investigational Site, Tokyo
  - GSK Investigational Site, Tottori
  - GSK Investigational Site, Yamagata

IPD SHARING:
Plan to Share IPD: Yes
Patient-level data for this study will be made available through www.clinicalstudydatarequest.com following the timelines and process described on this site.

REFERENCES:
- [Background] Tsukasa Koyama, Teruhiko Higuchi, Shigeto Yamawaki, Shigenobu Kanba, Takeshi Terao and Atsuko Shinohara. Study SCA106052, a clinical evaluation of BW430C (lamotrigine) in bipolar I disorder - Long-term extension study -. Rinsho seishin igaku. 2011;40(7):981-995.
- See also: Researchers can use this site to request access to anonymised patient level data and/or supporting documents from clinical studies to conduct further research. — https://www.clinicalstudydatarequest.com
- Available data/document: Individual Participant Data Set: SCA106052 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Annotated Case Report Form: SCA106052 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Statistical Analysis Plan: SCA106052 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Dataset Specification: SCA106052 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register

RESULTS

PARTICIPANT FLOW:
Groups:
- Lamotrigine - Dosage Adjustment Phase: Lamotrigine 12.5 milligrams per day (mg/day) to 200 mg/day for 6 weeks without any concomitant use of medication that induces lamotrigine glucuronidation
- Lamotrigine - Long-term Administration Phase: Lamotrigine 50 mg/day to 400 mg/day for 46 weeks depending on concomitant use of medication that induces or inhibits lamotrigine glucuronidation
Period: 6-week Dosage Adjustment Phase
Arm/Group | Lamotrigine - Dosage Adjustment Phase | Lamotrigine - Long-term Administration Phase
Started | 92 | 0
Completed | 85 | 0
Not Completed | 7 | 0
Not completed — Adverse Event | 5 | 0
Not completed — Lack of Efficacy | 2 | 0
Period: 46-week Long-term Administration Phase
Arm/Group | Lamotrigine - Dosage Adjustment Phase | Lamotrigine - Long-term Administration Phase
Started | 0 | 85
Completed | 0 | 68
Not Completed | 0 | 17
Not completed — Adverse Event | 0 | 7
Not completed — Physician Decision | 0 | 7
Not completed — Lost to Follow-up | 0 | 2
Not completed — Protocol-defined Stopping Criteria | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Lamotrigine: Dosage-adjustment Phase: lamotrigine 12.5 mg/day to 200 mg/day for 6 weeks without any concomitant use of medication that induces lamotrigine glucuronidation; followed by Long-term Administration Phase: lamotrigine 50 mg/day to 400 mg/day for 46 weeks depending on concomitant use of medication that induces or inhibits lamotrigine glucuronidation
Arm/Group | Lamotrigine
Number analyzed (Participants) | 92
Age, Continuous [Mean (Standard Deviation); unit: Years] | 43.5 (12.11)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 52
  Male | 40
Race/Ethnicity, Customized [Number; unit: participants]
  Asian - Japanese Heritage | 91
  Asian - East Asian Heritage | 1

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Any Serious Adverse Event (SAE) and Any Non Serious Adverse Event
Description: An adverse event (AE) is any untoward medical occurrence in a participant, temporally associated with the use of medicinal product, which does not necessarily have a causal relationship with the treatment. An SAE is any untoward medical occurrence that, at any dose, results in death, is life-threatening, requires inpatient hospitalization or causes its prolongation, results in persistent or significant disability/incapacity, is a congenital anomaly/birth defect, or is an important medical event. A complete list of all SAEs and AEs experienced in the study can be found in the SAE/AE section.
Time Frame: From baseline (Week 0) until 2 weeks after the end of treatment (Week 54)
Population: Safety Population: all participants who received at least one dose of study medication
Measure: Number; unit: participants
Groups:
- Lamotrigine: Dosage-adjustment Phase: lamotrigine 12.5 milligrams per day (mg/day) to 200 mg/day for 6 weeks without any concomitant use of medication that induces lamotrigine glucuronidation; followed by Long-term Administration Phase: lamotrigine 50 mg/day to 400 mg/day for 46 weeks depending on concomitant use of medication that induces or inhibits lamotrigine glucuronidation
Arm/Group | Lamotrigine
Number analyzed (Participants) | 92
participants
  Participants with any SAE | 13
  Participants with any non-serious AE | 75

2. Primary Outcome: Number of Participants With the Indicated Clinical Laboratory Test Values for Alkaline Phosphatase (ALP), Alanine Amino Transferase (ALT), Aspartate Amino Transferase (AST), Gamma Glutamyl Transferase (GGT), and Lactate Dehydrogenase (LDH)
Description: Participants in the study were evaluated for the following clinical laboratory parameters at the indicated time points: ALP, ALT, AST, GGT, and LDH. Participants were categorized as "High" for laboratory values above normal (reference) and as "Low" for laboratory values below normal ranges used by the central laboratory. Normal ranges: ALP, 104-338 International Units per liter (IU/L); ALT, 5-45 IU/L; AST, 10-40 IU/L; GGT, Male: 0-79 IU/L, Female: 0-48 IU/L; LDH 120-245 IU/L.
Time Frame: Baseline (Week 0) and Weeks 6, 16, 28, 40, and 52/Early Withdrawal (EW)
Population: Safety Population. The number of participants with an assessment varied depending on the number of assessments completed at each visit (indicated time points).
Measure: Number; unit: participants
Arm/Group | Lamotrigine
Number analyzed (Participants) | 92
participants
  ALP, High, Week 0; n=92 | 1
  ALP, Normal, Week 0; n=92 | 89
  ALP, Low, Week 0; n=92 | 2
  ALP, High, Week 6; n=84 | 2
  ALP, Normal, Week 6; n=84 | 82
  ALP, Low, Week 6; n=84 | 0
  ALP, High, Week 16; n=78 | 3
  ALP, Normal, Week 16; n=78 | 74
  ALP, Low, Week 16; n=78 | 1
  ALP, High, Week 28; n=77 | 1
  ALP, Normal, Week 28; n=77 | 76
  ALP, Low, Week 28; n=77 | 0
  ALP, High, Week 40; n=70 | 3
  ALP, Normal, Week 40; n=70 | 66
  ALP, Low, Week 40; n=70 | 1
  ALP, High, Week 52/EW; n=86 | 4
  ALP, Normal, Week 52/EW; n=86 | 81
  ALP, Low, Week 52/EW; n=86 | 1
  ALT, High, Week 0; n=92 | 6
  ALT, Normal, Week 0; n=92 | 86
  ALT, Low, Week 0; n=92 | 0
  ALT, High, Week 6; n=84 | 2
  ALT, Normal, Week 6; n=84 | 82
  ALT, Low, Week 6; n=84 | 0
  ALT, High, Week 16; n=78 | 3
  ALT, Normal, Week 16; n=78 | 75
  ALT, Low, Week 16; n=78 | 0
  ALT, High, Week 28; n=77 | 4
  ALT, Normal, Week 28; n=77 | 73
  ALT, Low, Week 28; n=77 | 0
  ALT, High, Week 40; n=70 | 3
  ALT, Normal, Week 40; n=70 | 67
  ALT, Low, Week 40; n=70 | 0
  ALT, High, Week 52/EW; n=86 | 3
  ALT, Normal, Week 52/EW; n=86 | 83
  ALT, Low, Week 52/EW; n=86 | 0
  AST, High, Week 0; n=92 | 3
  AST, Normal, Week 0; n=92 | 89
  AST, Low, Week 0; n=92 | 0
  AST, High, Week 6; n=84 | 2
  AST, Normal, Week 6; n=84 | 82
  AST, Low, Week 6; n=84 | 0
  AST, High, Week 16; n=78 | 2
  AST, Normal, Week 16; n=78 | 76
  AST, Low, Week 16; n=78 | 0
  AST, High, Week 28; n=77 | 2
  AST, Normal, Week 28; n=77 | 75
  AST, Low, Week 28; n=77 | 0
  AST, High, Week 40; n=70 | 3
  AST, Normal, Week 40; n=70 | 67
  AST, Low, Week 40; n=70 | 0
  AST, High, Week 52/EW; n=86 | 3
  AST, Normal, Week 52/EW; n=86 | 83
  AST, Low, Week 52/EW; n=86 | 0
  GGT, High, Week 0; n=92 | 5
  GGT, Normal, Week 0; n=92 | 87
  GGT, Low, Week 0; n=92 | 0
  GGT, High, Week 6; n=84 | 3
  GGT, Normal, Week 6; n=84 | 81
  GGT, Low, Week 6; n=84 | 0
  GGT, High, Week 16; n=78 | 4
  GGT, Normal, Week 16; n=78 | 74
  GGT, Low, Week 16; n=78 | 0
  GGT, High, Week 28; n=77 | 5
  GGT, Normal, Week 28; n=77 | 72
  GGT, Low, Week 28; n=77 | 0
  GGT, High, Week 40; n=70 | 4
  GGT, Normal, Week 40; n=70 | 66
  GGT, Low, Week 40; n=70 | 0
  GGT, High, Week 52/EW; n=86 | 5
  GGT, Normal, Week 52/EW; n=86 | 81
  GGT, Low, Week 52/EW; n=86 | 0
  LDH, High, Week 0; n=92 | 4
  LDH, Normal, Week 0; n=92 | 84
  LDH, Low, Week 0; n=92 | 4
  LDH, High, Week 6; n=84 | 4
  LDH, Normal, Week 6; n=84 | 77
  LDH, Low, Week 6; n=84 | 3
  LDH, High, Week 16; n=78 | 2
  LDH, Normal, Week 16; n=78 | 73
  LDH, Low, Week 16; n=78 | 3
  LDH, High, Week 28; n=77 | 3
  LDH, Normal, Week 28; n=77 | 72
  LDH, Low, Week 28; n=77 | 2
  LDH, High, Week 40; n=70 | 3
  LDH, Normal, Week 40; n=70 | 64
  LDH, Low, Week 40; n=70 | 3
  LDH, High, Week 52/EW; n=86 | 3
  LDH, Normal, Week 52/EW; n=86 | 82
  LDH, Low, Week 52/EW; n=86 | 1

3. Primary Outcome: Number of Participants With Clinical Laboratory Test Values Out of the Normal Range and in the Normal Range for Total Bilirubin and Creatinine at Weeks 0, 6, 16, 28, 40, and 52/EW
Description: Participants in the study were evaluated for the following clinical laboratory parameters at the indicated time points: total bilirubin and creatinine. Participants were categorized as "High" for laboratory values above normal (reference) and as "Low" for laboratory values below normal ranges used by the central laboratory. Normal ranges: total bilirubin, 3.42-17.1 micromoles per liter (UMOL/L); creatinine, Male: 57.46-96.356 UMOL/L, Female: 40.664-72.488 UMOL/L.
Time Frame: Baseline (Week 0) and Weeks 6, 16, 28, 40, and 52/EW
Population: as for outcome 2
Measure: Number; unit: participants
Arm/Group | Lamotrigine
Number analyzed (Participants) | 92
participants
  Total bilirubin, High, Week 0; n=92 | 5
  Total bilirubin, Normal, Week 0; n=92 | 87
  Total bilirubin, Low, Week 0; n=92 | 0
  Total bilirubin, High, Week 6; n=84 | 5
  Total bilirubin, Normal, Week 6; n=84 | 79
  Total bilirubin, Low, Week 6; n=84 | 0
  Total bilirubin, High, Week 16; n=78 | 2
  Total bilirubin, Normal, Week 16; n=78 | 76
  Total bilirubin, Low, Week 16; n=78 | 0
  Total bilirubin, High, Week 28; n=77 | 3
  Total bilirubin, Normal, Week 28; n=77 | 74
  Total bilirubin, Low, Week 28; n=77 | 0
  Total bilirubin, High, Week 40; n=70 | 4
  Total bilirubin, Normal, Week 40; n=70 | 66
  Total bilirubin, Low, Week 40; n=70 | 0
  Total bilirubin, High, Week 52/EW; n=86 | 8
  Total bilirubin, Normal, Week 52/EW; n=86 | 78
  Total bilirubin, Low, Week 52/EW; n=86 | 0
  Creatinine, High, Week 0; n=92 | 2
  Creatinine, Normal, Week 0; n=92 | 86
  Creatinine, Low, Week 0; n=92 | 4
  Creatinine, High, Week 6; n=84 | 2
  Creatinine, Normal, Week 6; n=84 | 81
  Creatinine, Low, Week 6; n=84 | 1
  Creatinine, High, Week 16; n=78 | 4
  Creatinine, Normal, Week 16; n=78 | 72
  Creatinine, Low, Week 16; n=78 | 2
  Creatinine, High, Week 28; n=77 | 2
  Creatinine, Normal, Week 28; n=77 | 73
  Creatinine, Low, Week 28; n=77 | 2
  Creatinine, High, Week 40; n=70 | 2
  Creatinine, Normal, Week 40; n=70 | 66
  Creatinine, Low, Week 40; n=70 | 2
  Creatinine, High, Week 52/EW; n=86 | 3
  Creatinine, Normal, Week 52/EW; n=86 | 79
  Creatinine, Low, Week 52/EW; n=86 | 4

4. Primary Outcome: Number of Participants With Clinical Laboratory Test Values Out of the Normal Range and in the Normal Range for Calcium, Cholesterol, Chloride, Potassium, Sodium, Triglycerides, and Urea/Blood Urea Nitrogen (BUN) at Weeks 0, 6, 16, 28, 40, and 52/EW
Description: Participants were evaluated for the following clinical laboratory parameters for blood chemistry at the indicated time points: electrolytes (calcium, chloride, potassium, sodium), cholesterol, triglycerides, and urea/BUN. Participants were categorized as "High" for laboratory values above normal (reference) and as "Low" for laboratory values below normal ranges used by the central laboratory. Normal ranges (micromoles per liter [MMOL/L]): calcium, 2.0459-2.495; chloride, 98-108; potassium, 3.5-5; sodium, 135-145; cholesterol, 3.879-5.66334; triglycerides, 0.565-1.6837; urea/BUN, 2.856-7.14.
Time Frame: Baseline (Week 0) and Weeks 6, 16, 28, 40, and 52/EW
Population: as for outcome 2
Measure: Number; unit: participants
Arm/Group | Lamotrigine
Number analyzed (Participants) | 92
participants
  Calcium, High, Week 0; n=92 | 1
  Calcium, Normal, Week 0; n=92 | 91
  Calcium, Low, Week 0; n=92 | 0
  Calcium, High, Week 6; n=84 | 4
  Calcium, Normal, Week 6; n=84 | 80
  Calcium, Low, Week 6; n=84 | 0
  Calcium, High, Week 16; n=78 | 2
  Calcium, Normal, Week 16; n=78 | 75
  Calcium, Low, Week 16; n=78 | 1
  Calcium, High, Week 28; n=77 | 1
  Calcium, Normal, Week 28; n=77 | 76
  Calcium, Low, Week 28; n=77 | 0
  Calcium, High, Week 40; n=70 | 1
  Calcium, Normal, Week 40; n=70 | 69
  Calcium, Low, Week 40; n=70 | 0
  Calcium, High, Week 52/EW; n=86 | 0
  Calcium, Normal, Week 52/EW; n=86 | 85
  Calcium, Low, Week 52/EW; n=86 | 1
  Cholesterol, High, Week 0; n=92 | 21
  Cholesterol, Normal, Week 0; n=92 | 66
  Cholesterol, Low, Week 0; n=92 | 5
  Cholesterol, High, Week 6; n=84 | 20
  Cholesterol, Normal, Week 6; n=84 | 57
  Cholesterol, Low, Week 6; n=84 | 7
  Cholesterol, High, Week 16; n=78 | 16
  Cholesterol, Normal, Week 16; n=78 | 58
  Cholesterol, Low, Week 16; n=78 | 4
  Cholesterol, High, Week 28; n=77 | 13
  Cholesterol, Normal, Week 28; n=77 | 61
  Cholesterol, Low, Week 28; n=77 | 3
  Cholesterol, High, Week 40; n=70 | 20
  Cholesterol, Normal, Week 40; n=70 | 45
  Cholesterol, Low, Week 40; n=70 | 5
  Cholesterol, High, Week 52/EW; n=86 | 18
  Cholesterol, Normal, Week 52/EW; n=86 | 64
  Cholesterol, Low, Week 52/EW; n=86 | 4
  Chloride, High, Week 0; n=92 | 2
  Chloride, Normal Week 0; n=92 | 90
  Chloride, Low, Week 0; n=92 | 0
  Chloride, High, Week 6; n=84 | 0
  Chloride, Normal, Week 6; n=84 | 84
  Chloride, Low, Week 6; n=84 | 0
  Chloride, High, Week 16; n=78 | 0
  Chloride, Normal, Week 16; n=78 | 77
  Chloride, Low, Week 16; n=78 | 1
  Chloride, High, Week 28; n=77 | 0
  Chloride, Normal, Week 28; n=77 | 76
  Chloride, Low, Week 28; n=77 | 1
  Chloride, High, Week 40; n=70 | 2
  Chloride, Normal, Week 40; n=70 | 66
  Chloride, Low, Week 40; n=70 | 2
  Chloride, High, Week 52/EW; n=86 | 3
  Chloride, Normal, Week 52/EW; n=86 | 79
  Chloride, Low, Week 52/EW; n=86 | 4
  Potassium, High, Week 0; n=92 | 0
  Potassium, Normal, Week 0; n=92 | 92
  Potassium, Low, Week 0; n=92 | 0
  Potassium, High, Week 6; n=84 | 1
  Potassium, Normal, Week 6; n=84 | 83
  Potassium, Low, Week 6; n=84 | 0
  Potassium, High, Week 16; n=78 | 2
  Potassium, Normal, Week 16; n=78 | 76
  Potassium, Low, Week 16; n=78 | 0
  Potassium, High, Week 28; n=77 | 0
  Potassium, Normal, Week 28; n=77 | 76
  Potassium, Low, Week 28; n=77 | 1
  Potassium, High, Week 40; n=70 | 2
  Potassium, Normal, Week 40; n=70 | 68
  Potassium, Low, Week 40; n=70 | 0
  Potassium, High, Week 52/EW; n=86 | 0
  Potassium, Normal, Week 52/EW; n=86 | 86
  Potassium, Low, Week 52/EW; n=86 | 0
  Sodium, High, Week 0; n=92 | 1
  Sodium, Normal, Week 0; n=92 | 90
  Sodium, Low, Week 0; n=92 | 1
  Sodium, High, Week 6; n=84 | 0
  Sodium, Normal, Week 6; n=84 | 83
  Sodium, Low, Week 6; n=84 | 1
  Sodium, High, Week 16; n=78 | 0
  Sodium, Normal, Week 16; n=78 | 77
  Sodium, Low, Week 16; n=78 | 1
  Sodium, High, Week 28; n=77 | 0
  Sodium, Normal, Week 28; n=77 | 76
  Sodium, Low, Week 28; n=77 | 1
  Sodium, High, Week 40; n=70 | 0
  Sodium, Normal, Week 40; n=70 | 69
  Sodium, Low, Week 40; n=70 | 1
  Sodium, High, Week 52/EW; n=86 | 1
  Sodium, Normal, Week 52/EW; n=86 | 83
  Sodium, Low, Week 52/EW; n=86 | 2
  Triglycerides, High, Week 0; n=92 | 23
  Triglycerides, Normal, Week 0; n=92 | 55
  Triglycerides, Low, Week 0; n=92 | 14
  Triglycerides, High, Week 6; n=84 | 20
  Triglycerides, Normal, Week 6; n=84 | 50
  Triglycerides, Low, Week 6; n=84 | 14
  Triglycerides, High, Week 16; n=78 | 20
  Triglycerides, Normal, Week 16; n=78 | 50
  Triglycerides, Low, Week 16; n=78 | 8
  Triglycerides, High, Week 28; n=77 | 23
  Triglycerides, Normal, Week 28; n=77 | 42
  Triglycerides, Low, Week 28; n=77 | 12
  Triglycerides, High, Week 40; n=70 | 18
  Triglycerides, Normal, Week 40; n=70 | 40
  Triglycerides, Low, Week 40; n=70 | 12
  Triglycerides, High, Week 52/EW; n=86 | 21
  Triglycerides, Normal, Week 52/EW; n=86 | 53
  Triglycerides, Low, Week 52/EW; n=86 | 12
  Urea/BUN, High, Week 0; n=92 | 4
  Urea/BUN, Normal, Week 0; n=92 | 77
  Urea/BUN, Low, Week 0; n=92 | 11
  Urea/BUN, High, Week 6; n=84 | 1
  Urea/BUN, Normal, Week 6; n=84 | 74
  Urea/BUN, Low, Week 6; n=84 | 9
  Urea/BUN, High, Week 16; n=78 | 5
  Urea/BUN, Normal, Week 16; n=78 | 68
  Urea/BUN, Low, Week 16; n=78 | 5
  Urea/BUN, High, Week 28; n=77 | 2
  Urea/BUN, Normal, Week 28; n=77 | 73
  Urea/BUN, Low, Week 28; n=77 | 2
  Urea/BUN, High, Week 40; n=70 | 5
  Urea/BUN, Normal, Week 40; n=70 | 56
  Urea/BUN, Low, Week 40; n=70 | 9
  Urea/BUN, High, Week 52/EW; n=86 | 5
  Urea/BUN, Normal, Week 52/EW; n=86 | 74
  Urea/BUN, Low, Week 52/EW; n=86 | 7

5. Primary Outcome: Number of Participants With Clinical Laboratory Test Values Out of the Normal Range and in the Normal Range for Platelet Count and White Blood Cell Count at Weeks 0, 6, 16, 28, 40, and 52/EW
Description: Participants in the study were evaluated for the following clinical laboratory parameters of hematology at the indicated time points: platelet count and white blood cell count. Participants were categorized as "High" for laboratory values above normal (reference) and as "Low" for laboratory values below normal ranges used by the central laboratory. Normal ranges: platelet count, 140-379 GI (gibi; 10^9) per liter (GI/L); white blood cell count, 3.5-9.7 GI/L.
Time Frame: Baseline (Week 0) and Weeks 6, 16, 28, 40, and 52/EW
Population: as for outcome 2
Measure: Number; unit: participants
Arm/Group | Lamotrigine
Number analyzed (Participants) | 92
participants
  Platelet count, High, Week 0; n=92 | 3
  Platelet count, Normal, Week 0; n=92 | 89
  Platelet count, Low, Week 0; n=92 | 0
  Platelet count, High, Week 6; n=84 | 2
  Platelet count, Normal, Week 6; n=84 | 81
  Platelet count, Low, Week 6; n=84 | 1
  Platelet count, High, Week 16; n=78 | 2
  Platelet count, Normal, Week 16; n=78 | 75
  Platelet count, Low, Week 16; n=78 | 1
  Platelet count, High, Week 28; n=77 | 2
  Platelet count, Normal, Week 28; n=77 | 75
  Platelet count, Low, Week 28; n=77 | 0
  Platelet count, High, Week 40; n=68 | 0
  Platelet count, Normal, Week 40; n=68 | 68
  Platelet count, Low, Week 40; n=68 | 0
  Platelet count, High, Week 52/EW; n=86 | 3
  Platelet count, Normal, Week 52/EW; n=86 | 82
  Platelet count, Low, Week 52/EW; n=86 | 1
  White blood cell count, High, Week 0; n=92 | 7
  White blood cell count, Normal, Week 0; n=92 | 83
  White blood cell count, Low, Week 0; n=92 | 2
  White blood cell count, High, Week 6; n=84 | 1
  White blood cell count, Normal, Week 6; n=84 | 81
  White blood cell count, Low, Week 6; n=84 | 2
  White blood cell count, High, Week 16; n=78 | 1
  White blood cell count, Normal, Week 16; n=78 | 75
  White blood cell count, Low, Week 16; n=78 | 2
  White blood cell count, High, Week 28; n=77 | 2
  White blood cell count, Normal, Week 28; n=77 | 70
  White blood cell count, Low, Week 28; n=77 | 5
  White blood cell count, High, Week 40; n=69 | 3
  White blood cell count, Normal, Week 40; n=69 | 61
  White blood cell count, Low, Week 40; n=69 | 5
  White blood cell count, High, Week 52/EW; n=86 | 3
  White blood cell count, Normal, Week 52/EW; n=86 | 80
  White blood cell count, Low, Week 52/EW; n=86 | 3

6. Primary Outcome: Number of Participants With Clinical Laboratory Test Values Out of the Normal Range and in the Normal Range for Total Protein, Hemoglobin, and Hematocrit at Weeks 0, 6, 16, 28, 40, and 52/EW
Description: Participants in the study were evaluated for total protein, hemoglobin, and hematocrit at the indicated time points. Participants were categorized as "High" for laboratory values above normal (reference) and as "Low" for laboratory values below normal ranges used by the central laboratory. Normal ranges: total protein, 65-82 grams per liter (G/L); hemoglobin, Male: 136-183 G/L, Female: 112-152 G/L; hematocrit (proportion of 1), Male: 0.404-0.519, Female: 0.343-0.452.
Time Frame: Baseline (Week 0) and Weeks 6, 16, 28, 40, and 52/EW
Population: as for outcome 2
Measure: Number; unit: participants
Arm/Group | Lamotrigine
Number analyzed (Participants) | 92
participants
  Total protein, High, Week 0; n=92 | 1
  Total protein, Normal, Week 0; n=92 | 85
  Total protein, Low, Week 0; n=92 | 6
  Total protein, High, Week 6; n=84 | 0
  Total protein, Normal, Week 6; n=84 | 77
  Total protein, Low, Week 6; n=84 | 7
  Total protein, High, Week 16; n=78 | 0
  Total protein, Normal, Week 16; n=78 | 74
  Total protein, Low, Week 16; n=78 | 4
  Total protein, High, Week 28; n=77 | 0
  Total protein, Normal, Week 28; n=77 | 69
  Total protein, Low, Week 28; n=77 | 8
  Total protein, High, Week 40; n=70 | 1
  Total protein, Normal, Week 40; n=70 | 64
  Total protein, Low, Week 40; n=70 | 5
  Total protein, High, Week 52/EW; n=86 | 0
  Total protein, Normal, Week 52/EW; n=86 | 72
  Total protein, Low, Week 52/EW; n=86 | 14
  Hemoglobin, High, Week 0; n=92 | 4
  Hemoglobin, Normal, Week 0; n=92 | 80
  Hemoglobin, Low, Week 0; n=92 | 8
  Hemoglobin, High, Week 6; n=84 | 2
  Hemoglobin, Normal, Week 6; n=84 | 75
  Hemoglobin, Low, Week 6; n=84 | 7
  Hemoglobin, High, Week 16; n=78 | 3
  Hemoglobin, Normal, Week 16; n=78 | 68
  Hemoglobin, Low, Week 16; n=78 | 7
  Hemoglobin, High, Week 28; n=77 | 1
  Hemoglobin, Normal, Week 28; n=77 | 69
  Hemoglobin, Low, Week 28; n=77 | 7
  Hemoglobin, High, Week 40; n=69 | 1
  Hemoglobin, Normal, Week 40; n=69 | 62
  Hemoglobin, Low, Week 40; n=69 | 6
  Hemoglobin, High, Week 52/EW; n=86 | 4
  Hemoglobin, Normal, Week 52/EW; n=86 | 71
  Hemoglobin, Low, Week 52/EW; n=86 | 11
  Hematocrit, High, Week 0; n=92 | 4
  Hematocrit, Normal, Week 0; n=92 | 83
  Hematocrit, Low, Week 0; n=92 | 5
  Hematocrit, High, Week 6; n=84 | 3
  Hematocrit, Normal, Week 6; n=84 | 75
  Hematocrit, Low, Week 6; n=84 | 6
  Hematocrit, High, Week 16; n=78 | 2
  Hematocrit, Normal, Week 16; n=78 | 73
  Hematocrit, Low, Week 16; n=78 | 3
  Hematocrit, High, Week 28; n=77 | 3
  Hematocrit, Normal, Week 28; n=77 | 69
  Hematocrit, Low, Week 28; n=77 | 5
  Hematocrit, High, Week 40; n=69 | 4
  Hematocrit, Normal, Week 40; n=69 | 63
  Hematocrit, Low, Week 40; n=69 | 2
  Hematocrit, High, Week 52/EW; n=86 | 3
  Hematocrit, Normal, Week 52/EW; n=86 | 73
  Hematocrit, Low, Week 52/EW; n=86 | 10

7. Primary Outcome: Number of Participants With Clinical Laboratory Test Values Out of the Normal Range and in the Normal Range for Red Blood Cell Count at Weeks 0, 6, 16, 28, 40, and 52/EW
Description: Red blood cell count was measured in participants at the indicated time points. Participants were categorized as "High" for laboratory values above normal (reference) and as "Low" for laboratory values below normal ranges used by the central laboratory. Normal ranges: red blood cell count, Male: 4.38-5.77 TI (tebi; 10^12)/L, Female: 3.76-5.16 TI/L.
Time Frame: Baseline (Week 0) and Weeks 6, 16, 28, 40, and 52/EW
Population: as for outcome 2
Measure: Number; unit: participants
Arm/Group | Lamotrigine
Number analyzed (Participants) | 92
participants
  Red blood cell count, High, Week 0; n=92 | 2
  Red blood cell count, Normal, Week 0; n=92 | 88
  Red blood cell count, Low, Week 0; n=92 | 2
  Red blood cell count, High, Week 6; n=84 | 1
  Red blood cell count, Normal, Week 6; n=84 | 78
  Red blood cell count, Low, Week 6; n=84 | 5
  Red blood cell count, High, Week 16; n=78 | 1
  Red blood cell count, Normal, Week 16; n=78 | 73
  Red blood cell count, Low, Week 16; n=78 | 4
  Red blood cell count, High, Week 28; n=77 | 1
  Red blood cell count, Normal, Week 28; n=77 | 70
  Red blood cell count, Low, Week 28; n=77 | 6
  Red blood cell count, High, Week 40; n=69 | 1
  Red blood cell count, Normal, Week 40; n=69 | 64
  Red blood cell count, Low, Week 40; n=69 | 4
  Red blood cell count, High, Week 52/EW; n=86 | 3
  Red blood cell count, Normal, Week 52/EW; n=86 | 72
  Red blood cell count, Low, Week 52/EW; n=86 | 11

8. Primary Outcome: Number of Participants in the Indicated Category for Urine Glucose, Urine Protein, and Urine Urobilinogen at Baseline (Week 0) and Weeks 6, 16, 28, 40, and 52/EW
Description: Urine glucose, urine protein, and urine urobilinogen were measured in participants at the indicated time points. In this dipstick (qualitative) test, the level of glucose, protein, and urobilinogen in urine samples was recorded as negative (NEG [-]), trace (TRA [+/-]), 1+, 2+, 3+, 4+, and 5+ (the plus sign increases with a higher level of glucose, protein, or urobilinogen in the urine: 1+=slightly positive, 2+=positive, 3+=high positive, 4+=very high positive, 5+=more positive than 4+).
Time Frame: Baseline (Week 0) and Weeks 6, 16, 28, 40, and 52/EW
Population: as for outcome 2
Measure: Number; unit: participants
Arm/Group | Lamotrigine
Number analyzed (Participants) | 92
participants
  Urine Glucose, Week 0, NEG [-]; n=92 | 88
  Urine Glucose, Week 0, TRA [+/-]; n=92 | 1
  Urine Glucose, Week 0, 1+; n=92 | 1
  Urine Glucose, Week 0, 2+; n=92 | 1
  Urine Glucose, Week 0, 3+; n=92 | 0
  Urine Glucose, Week 0, 4+; n=92 | 1
  Urine Glucose, Week 0, 5+; n=92 | 0
  Urine Glucose, Week 6, NEG [-]; n=84 | 81
  Urine Glucose, Week 6, TRA [+/-]; n=84 | 0
  Urine Glucose, Week 6, 1+; n=84 | 1
  Urine Glucose, Week 6, 2+; n=84 | 1
  Urine Glucose, Week 6, 3+; n=84 | 1
  Urine Glucose, Week 6, 4+; n=84 | 0
  Urine Glucose, Week 6, 5+; n=84 | 0
  Urine Glucose, Week 16, NEG [-]; n=78 | 77
  Urine Glucose, Week 16, TRA [+/-]; n=78 | 0
  Urine Glucose, Week 16, 1+; n=78 | 1
  Urine Glucose, Week 16, 2+; n=78 | 0
  Urine Glucose, Week 16, 3+; n=78 | 0
  Urine Glucose, Week 16, 4+; n=78 | 0
  Urine Glucose, Week 16, 5+; n=78 | 0
  Urine Glucose, Week 28, NEG [-]; n=77 | 76
  Urine Glucose, Week 28, TRA [+/-]; n=77 | 1
  Urine Glucose, Week 28, 1+; n=77 | 0
  Urine Glucose, Week 28, 2+; n=77 | 0
  Urine Glucose, Week 28, 3+; n=77 | 0
  Urine Glucose, Week 28, 4+; n=77 | 0
  Urine Glucose, Week 28, 5+; n=77 | 0
  Urine Glucose, Week 40, NEG [-]; n=70 | 68
  Urine Glucose, Week 40, TRA [+/-]; n=70 | 2
  Urine Glucose, Week 40, 1+; n=70 | 0
  Urine Glucose, Week 40, 2+; n=70 | 0
  Urine Glucose, Week 40, 3+; n=70 | 0
  Urine Glucose, Week 40, 4+; n=70 | 0
  Urine Glucose, Week 40, 5+; n=70 | 0
  Urine Glucose, Week 52/EW, NEG [-]; n=86 | 85
  Urine Glucose, Week 52/EW, TRA [+/-]; n=86 | 0
  Urine Glucose, Week 52/EW, 1+; n=86 | 1
  Urine Glucose, Week 52/EW, 2+; n=86 | 0
  Urine Glucose, Week 52/EW, 3+; n=86 | 0
  Urine Glucose, Week 52/EW, 4+; n=86 | 0
  Urine Glucose, Week 52/EW, 5+; n=86 | 0
  Urine Protein, Week 0, NEG [-]; n=92 | 87
  Urine Protein, Week 0, TRA [+/-]; n=92 | 3
  Urine Protein, Week 0, 1+; n=92 | 1
  Urine Protein, Week 0, 2+; n=92 | 1
  Urine Protein, Week 0, 3+; n=92 | 0
  Urine Protein, Week 0, 4+; n=92 | 0
  Urine Protein, Week 0, 5+; n=92 | 0
  Urine Protein, Week 6, NEG [-]; n=84 | 81
  Urine Protein, Week 6, TRA [+/-]; n=84 | 1
  Urine Protein, Week 6, 1+; n=84 | 2
  Urine Protein, Week 6, 2+; n=84 | 0
  Urine Protein, Week 6, 3+; n=84 | 0
  Urine Protein, Week 6, 4+; n=84 | 0
  Urine Protein, Week 6, 5+; n=84 | 0
  Urine Protein, Week 16, NEG [-]; n=78 | 76
  Urine Protein, Week 16, TRA [+/-]; n=78 | 0
  Urine Protein, Week 16, 1+; n=78 | 1
  Urine Protein, Week 16, 2+; n=78 | 1
  Urine Protein, Week 16, 3+; n=78 | 0
  Urine Protein, Week 16, 4+; n=78 | 0
  Urine Protein, Week 16, 5+; n=78 | 0
  Urine Protein, Week 28, NEG [-]; n=77 | 75
  Urine Protein, Week 28, TRA [+/-]; n=77 | 0
  Urine Protein, Week 28, 1+; n=77 | 2
  Urine Protein, Week 28, 2+; n=77 | 0
  Urine Protein, Week 28, 3+; n=77 | 0
  Urine Protein, Week 28, 4+; n=77 | 0
  Urine Protein, Week 28, 5+; n=77 | 0
  Urine Protein, Week 40, NEG [-]; n=70 | 69
  Urine Protein, Week 40, TRA [+/-]; n=70 | 0
  Urine Protein, Week 40, 1+; n=70 | 0
  Urine Protein, Week 40, 2+; n=70 | 1
  Urine Protein, Week 40, 3+; n=70 | 0
  Urine Protein, Week 40, 4+; n=70 | 0
  Urine Protein, Week 40, 5+; n=70 | 0
  Urine Protein, Week 52/EW, NEG [-]; n=86 | 81
  Urine Protein, Week 52/EW, TRA [+/-]; n=86 | 1
  Urine Protein, Week 52/EW, 1+; n=86 | 3
  Urine Protein, Week 52/EW, 2+; n=86 | 1
  Urine Protein, Week 52/EW, 3+; n=86 | 0
  Urine Protein, Week 52/EW, 4+; n=86 | 0
  Urine Protein, Week 52/EW, 5+; n=86 | 0
  Urine Urobilinogen, Week 0, NEG [-]; n=92 | 0
  Urine Urobilinogen, Week 0, TRA [+/-]; n=92 | 88
  Urine Urobilinogen, Week 0, 1+; n=92 | 4
  Urine Urobilinogen, Week 0, 2+; n=92 | 0
  Urine Urobilinogen, Week 0, 3+; n=92 | 0
  Urine Urobilinogen, Week 0, 4+; n=92 | 0
  Urine Urobilinogen, Week 0, 5+; n=92 | 0
  Urine Urobilinogen, Week 6, NEG [-]; n=84 | 0
  Urine Urobilinogen, Week 6, TRA [+/-]; n=84 | 81
  Urine Urobilinogen, Week 6, 1+; n=84 | 2
  Urine Urobilinogen, Week 6, 2+; n=84 | 1
  Urine Urobilinogen, Week 6, 3+; n=84 | 0
  Urine Urobilinogen, Week 6, 4+; n=84 | 0
  Urine Urobilinogen, Week 6, 5+; n=84 | 0
  Urine Urobilinogen, Week 16, NEG [-]; n=78 | 0
  Urine Urobilinogen, Week 16, TRA [+/-]; n=78 | 76
  Urine Urobilinogen, Week 16, 1+; n=78 | 2
  Urine Urobilinogen, Week 16, 2+; n=78 | 0
  Urine Urobilinogen, Week 16, 3+; n=78 | 0
  Urine Urobilinogen, Week 16, 4+; n=78 | 0
  Urine Urobilinogen, Week 16, 5+; n=78 | 0
  Urine Urobilinogen, Week 28, NEG [-]; n=77 | 0
  Urine Urobilinogen, Week 28, TRA [+/-]; n=77 | 77
  Urine Urobilinogen, Week 28, 1+; n=77 | 0
  Urine Urobilinogen, Week 28, 2+; n=77 | 0
  Urine Urobilinogen, Week 28, 3+; n=77 | 0
  Urine Urobilinogen, Week 28, 4+; n=77 | 0
  Urine Urobilinogen, Week 28, 5+; n=77 | 0
  Urine Urobilinogen, Week 40, NEG [-]; n=70 | 0
  Urine Urobilinogen, Week 40, TRA [+/-]; n=70 | 68
  Urine Urobilinogen, Week 40, 1+; n=70 | 2
  Urine Urobilinogen, Week 40, 2+; n=70 | 0
  Urine Urobilinogen, Week 40, 3+; n=70 | 0
  Urine Urobilinogen, Week 40, 4+; n=70 | 0
  Urine Urobilinogen, Week 40, 5+; n=70 | 0
  Urine Urobilinogen, Week 52/EW, NEG [-]; n=86 | 0
  Urine Urobilinogen, Week 52/EW, TRA [+/-]; n=86 | 82
  Urine Urobilinogen, Week 52/EW, 1+; n=86 | 4
  Urine Urobilinogen, Week 52/EW, 2+; n=86 | 0
  Urine Urobilinogen, Week 52/EW, 3+; n=86 | 0
  Urine Urobilinogen, Week 52/EW, 4+; n=86 | 0
  Urine Urobilinogen, Week 52/EW, 5+; n=86 | 0

9. Primary Outcome: Mean Systolic Blood Pressure and Diastolic Blood Pressure of Participants at Baseline (Week 0) and Weeks 2, 4, 5, 6, 8, 12, 16, 20, 24, 28, 32, 36, 40, 44, 48, and 52/EW
Description: Systolic and diastolic blood pressure was measured in participants at the indicated time points.
Time Frame: Baseline (Week 0) and Weeks 2, 4, 5, 6, 8, 12, 16, 20, 24, 28, 32, 36, 40, 44, 48, and 52/EW
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Millimeters of mercury
Arm/Group | Lamotrigine
Number analyzed (Participants) | 92
Millimeters of mercury
  Systolic blood pressure, Week 0; n=92 | 119.9 (15.40)
  Systolic blood pressure, Week 2; n=87 | 121.7 (16.11)
  Systolic blood pressure, Week 4; n=85 | 118.9 (15.77)
  Systolic blood pressure, Week 5; n=85 | 119.0 (16.26)
  Systolic blood pressure, Week 6; n=84 | 120.4 (16.09)
  Systolic blood pressure, Week 8; n=81 | 118.6 (16.28)
  Systolic blood pressure, Week 12; n=79 | 120.1 (15.71)
  Systolic blood pressure, Week 16; n=78 | 119.1 (16.76)
  Systolic blood pressure, Week 20; n=77 | 117.8 (15.04)
  Systolic blood pressure, Week 24; n=77 | 118.5 (15.30)
  Systolic blood pressure, Week 28; n=77 | 117.3 (18.84)
  Systolic blood pressure, Week 32; n=76 | 121.8 (17.04)
  Systolic blood pressure, Week 36; n=73 | 121.3 (15.80)
  Systolic blood pressure, Week 40; n=70 | 118.2 (15.21)
  Systolic blood pressure, Week 44; n=69 | 118.7 (14.88)
  Systolic blood pressure, Week 48; n=69 | 121.2 (16.37)
  Systolic blood pressure, Week 52/EW; n=87 | 118.2 (14.20)
  Diastolic blood pressure, Week 0; n=92 | 74.2 (11.41)
  Diastolic blood pressure, Week 2; n=87 | 74.9 (11.62)
  Diastolic blood pressure, Week 4; n=85 | 74.2 (12.08)
  Diastolic blood pressure, Week 5; n=85 | 73.8 (12.34)
  Diastolic blood pressure, Week 6; n=84 | 73.7 (11.16)
  Diastolic blood pressure, Week 8; n=81 | 72.6 (12.72)
  Diastolic blood pressure, Week 12; n=79 | 73.2 (12.08)
  Diastolic blood pressure, Week 16; n=78 | 73.0 (12.29)
  Diastolic blood pressure, Week 20; n=77 | 73.6 (11.59)
  Diastolic blood pressure, Week 24; n=77 | 74.2 (11.72)
  Diastolic blood pressure, Week 28; n=77 | 71.1 (12.24)
  Diastolic blood pressure, Week 32; n=76 | 74.0 (11.93)
  Diastolic blood pressure, Week 36; n=73 | 72.4 (10.98)
  Diastolic blood pressure, Week 40; n=70 | 72.3 (12.04)
  Diastolic blood pressure, Week 44; n=69 | 73.0 (12.22)
  Diastolic blood pressure, Week 48; n=69 | 72.7 (11.91)
  Diastolic blood pressure, Week 52/EW; n=87 | 73.2 (11.69)

10. Primary Outcome: Mean Heart Rate of Participants at Week 0 (Baseline) and Weeks 2, 4, 5, 6, 8, 12, 16, 20, 24, 28, 32, 36, 40, 44, 48, and 52/EW
Description: Heart rate was measured in participants at the indicated time points.
Time Frame: Baseline (Week 0) and Weeks 2, 4, 5, 6, 8, 12, 16, 20, 24, 28, 32, 36, 40, 44, 48, and 52/EW
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: beat per minute
Arm/Group | Lamotrigine
Number analyzed (Participants) | 92
beat per minute
  Week 0; n=92 | 76.3 (12.48)
  Week 2; n=87 | 78.0 (12.77)
  Week 4; n=85 | 77.4 (11.96)
  Week 5; n=85 | 78.5 (12.54)
  Week 6; n=84 | 77.0 (11.97)
  Week 8; n=81 | 76.8 (11.34)
  Week 12; n=79 | 79.0 (13.47)
  Week 16; n=78 | 76.5 (11.81)
  Week 20; n=77 | 77.4 (11.09)
  Week 24; n=77 | 74.9 (12.50)
  Week 28; n=77 | 75.9 (10.28)
  Week 32; n=76 | 77.2 (12.23)
  Week 36; n=73 | 76.8 (11.46)
  Week 40; n=70 | 75.8 (10.63)
  Week 44; n=69 | 77.3 (11.10)
  Week 48; n=69 | 78.2 (11.63)
  Week 52/EW; n=87 | 74.8 (11.75)

11. Primary Outcome: Mean Weight of Participants at Baseline (Week 0) and Weeks 6, 8, 12, 16, 20, 24, 28, 32, 36, 40, 44, 48, and 52/EW
Description: The weight of participants was recorded at the indicated time points.
Time Frame: Baseline (Week 0) and Weeks 6, 8, 12, 16, 20, 24, 28, 32, 36, 40, 44, 48, and 52/EW
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: kilograms
Arm/Group | Lamotrigine
Number analyzed (Participants) | 92
kilograms
  Week 0; n=92 | 60.86 (12.532)
  Week 6; n=84 | 61.62 (12.405)
  Week 8; n=81 | 61.29 (12.420)
  Week 12; n=79 | 61.26 (12.685)
  Week 16; n=78 | 61.38 (12.753)
  Week 20; n=77 | 61.19 (12.929)
  Week 24; n=77 | 61.29 (12.712)
  Week 28; n=77 | 60.99 (12.688)
  Week 32; n=76 | 61.05 (12.840)
  Week 36; n=73 | 61.06 (13.097)
  Week 40; n=70 | 60.67 (13.214)
  Week 44; n=69 | 60.72 (13.214)
  Week 48; n=69 | 60.43 (13.056)
  Week 52/EW; n=87 | 60.09 (12.765)

12. Primary Outcome: Mean Body Mass Index (BMI) of All Participants at Week 0 (Baseline) and Weeks 6, 8, 12, 16, 20, 24, 28, 32,36, 40, 44, 48, and 52/EW
Description: The BMI for participants was calculated at the indicated time points as body weight in kilograms divided by height in meters squared.
Time Frame: Baseline (Week 0) and Weeks 0, 6, 8, 12, 16, 20, 24, 28, 32, 36, 40, 44, 48, and 52/EW
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Kilograms per meters squared
Arm/Group | Lamotrigine
Number analyzed (Participants) | 92
Kilograms per meters squared
  Week 0; n=92 | 22.8 (3.934)
  Week 6; n=84 | 23.01 (3.878)
  Week 8; n=81 | 22.89 (3.863)
  Week 12; n=79 | 22.93 (3.975)
  Week 16; n=78 | 22.96 (3.965)
  Week 20; n=77 | 22.86 (3.941)
  Week 24; n=77 | 22.91 (3.916)
  Week 28; n=77 | 22.80 (3.970)
  Week 32; n=76 | 22.81 (4.016)
  Week 36; n=73 | 22.71 (4.041)
  Week 40; n=70 | 22.48 (3.820)
  Week 44; n=69 | 22.51 (3.785)
  Week 48; n=69 | 22.40 (3.750)
  Week 52/EW; n=87 | 22.42 (3.818)

13. Primary Outcome: Number of Participants With the Indicated Electrocardiogram (ECG) Findings at Weeks 0, 6, 28, and 52/EW
Description: ECGs were recorded in participants at the indicated time points. ECG findings, as determined by the physicians, were reported as normal, abnormal but not clinically significant (NCS), abnormal but clinically significant (CS), and no result. Specific definitions of ECG categorizations were not provided; physicians were expected to apply reasonable standards of clinical judgment.
Time Frame: Weeks 0, 6, 28, and 52/EW
Population: as for outcome 2
Measure: Number; unit: participants
Arm/Group | Lamotrigine
Number analyzed (Participants) | 92
participants
  Week 0, Normal; n=92 | 73
  Week 0, Abnormal-NCS; n=92 | 19
  Week 0, Abnormal-CS; n=92 | 0
  Week 0, No result; n=92 | 0
  Week 6, Normal; n=84 | 69
  Week 6, Abnormal-NCS; n=84 | 15
  Week 6, Abnormal-CS; n=84 | 0
  Week 6, No result; n=84 | 0
  Week 28, Normal; n=77 | 62
  Week 28, Abnormal-NCS; n=77 | 15
  Week 28, Abnormal-CS; n=77 | 0
  Week 28, No result; n=77 | 0
  Week 52 (EW), Normal; n=84 | 68
  Week 52 (EW), Abnormal-NCS; n=84 | 15
  Week 52 (EW), Abnormal-CS; n=84 | 1
  Week 52 (EW), No result; n=84 | 0

14. Secondary Outcome: Clinical Global Impressions of Severity (CGI-S) Total Score at Weeks 0, 2, 4, 5, 6, 8, 12, 16, 20, 24, 28, 32, 36, 40, 44, 48, and 52/EW
Description: The CGI-S is a standardized assessment tool that uses a 7-point scale to assess a participant's severity of illness. The total score ranges from 0 to 7: 0=not assessed, 1=normal, 2=borderline ill, 3=mildly ill, 4=moderately ill, 5=markedly ill, 6=severly ill, 7=extremely ill. Higher scores reflect a higher severity of current illness states. The number of participants with an assessment varied depending on the number of assessments completed at each visit (indicated time points).
Time Frame: Weeks 0, 2, 4, 5, 6, 8, 12, 16, 20, 24, 28, 32, 36, 40, 44, 48, and 52/EW
Population: Full Analysis Set (FAS): participants who received >=1 dose of study medication and underwent >=1 efficacy assessment. Observed Cases (OC; observed data with no imputation) and Last Observation Carried Forward (LOCF; data imputed [replaced] by most recent observed value [compared to planned date of missing observation]) were used for analysis.
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Lamotrigine
Number analyzed (Participants) | 92
scores on a scale
  Week 0, LOCF; n=92 | 2.9 (1.10)
  Week 0, OC; n=92 | 2.9 (1.10)
  Week 2, LOCF; n=91 | 2.6 (1.19)
  Week 2, OC; n=87 | 2.5 (1.13)
  Week 4, LOCF; n=92 | 2.5 (1.17)
  Week 4, OC; n=85 | 2.3 (0.98)
  Week 5, LOCF; n=92 | 2.4 (1.16)
  Week 5, OC; n=85 | 2.2 (0.95)
  Week 6, LOCF; n=92 | 2.3 (1.13)
  Week 6, OC; n=84 | 2.2 (0.89)
  Week 8, LOCF; n=92 | 2.4 (1.16)
  Week 8, OC; n=81 | 2.2 (0.93)
  Week 12, LOCF; n=92 | 2.2 (1.20)
  Week 12, OC; n=79 | 2.0 (0.91)
  Week 16, LOCF; n=92 | 2.3 (1.21)
  Week 16, OC; n=78 | 2.1 (0.94)
  Week 20, LOCF; n=92 | 2.4 (1.22)
  Week 20, OC; n=77 | 2.1 (0.96)
  Week 24, LOCF; n=92 | 2.4 (1.20)
  Week 24, OC; n=77 | 2.2 (0.95)
  Week 28, LOCF; n=92 | 2.3 (1.24)
  Week 28, OC; n=77 | 2.1 (0.99)
  Week 32, LOCF; n=92 | 2.4 (1.19)
  Week 32, OC; n=76 | 2.2 (0.93)
  Week 36, LOCF; n=92 | 2.3 (1.23)
  Week 36, OC; n=73 | 2.0 (0.95)
  Week 40, LOCF; n=92 | 2.4 (1.22)
  Week 40, OC; n=70 | 2.1 (0.95)
  Week 44, LOCF; n=92 | 2.4 (1.23)
  Week 44, OC; n=69 | 2.1 (0.93)
  Week 48, LOCF; n=92 | 2.3 (1.23)
  Week 48, OC; n=69 | 2.0 (0.91)
  Week 52/EW, LOCF; n=92 | 2.1 (1.24)
  Week 52/EW, OC; n=87 | 2.1 (1.25)

15. Secondary Outcome: Change From Baseline in the Clinical Global Impressions of Severity (CGI-S) Total Score at Weeks 2, 4, 5, 6, 8, 12, 16, 20, 24, 28, 32, 36, 40, 44, 48, and 52/EW
Description: The CGI-S is a standardized assessment tool that uses a 7-point scale to assess a participant's severity of illness. The total score ranges from 0 to 7: 0=not assessed, 1=normal, 2=borderline ill, 3=mildly ill, 4=moderately ill, 5=markedly ill, 6=severly ill, 7=extremely ill. Higher scores reflect a higher severity of current illness states. Change from baseline was calculated as the values at Weeks 2, 4, 5, 6, 8, 12, 16, 20, 24, 28, 32, 36, 40, 44, 48 and 52 (or EW) minus the baseline value (Week 0).
Time Frame: Baseline (Week 0) and Weeks 2, 4, 5, 6, 8, 12, 16, 20, 24, 28, 32, 36, 40, 44, 48, and 52/EW
Population: FAS Population. OC and LOCF datasets were used for analysis. The number of participants with an assessment varied depending on the number of assessments completed at each visit (indicated time points).
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Lamotrigine
Number analyzed (Participants) | 92
scores on a scale
  Week 2, LOCF; n=91 | -0.3 (0.93)
  Week 2, OC; n=87 | -0.3 (0.92)
  Week 4, LOCF; n=92 | -0.4 (1.01)
  Week 4, OC; n=85 | -0.5 (0.96)
  Week 5, LOCF; n=92 | -0.5 (1.07)
  Week 5, LOCF; n=85 | -0.6 (1.03)
  Week 6, LOCF; n=92 | -0.6 (1.07)
  Week 6, OC; n=84 | -0.7 (1.02)
  Week 8, LOCF; n=92 | -0.5 (1.16)
  Week 8, LOCF; n=81 | -0.6 (1.14)
  Week 12, LOCF; n=92 | -0.7 (1.23)
  Week 12, OC; n=79 | -0.8 (1.19)
  Week 16, LOCF; n=92 | -0.6 (1.21)
  Week 16, OC; n=78 | -0.7 (1.17)
  Week 20, LOCF; n=92 | -0.5 (1.17)
  Week 20, OC; n=77 | -0.6 (1.14)
  Week 24, LOCF; n=92 | -0.5 (1.09)
  Week 24, OC; n=77 | -0.6 (1.05)
  Week 28, LOCF; n=92 | -0.5 (1.23)
  Week 28, OC; n=77 | -0.7 (1.21)
  Week 32, LOCF; n=92 | -0.5 (1.14)
  Week 32, OC; n=76 | -0.6 (1.11)
  Week 36, LOCF; n=92 | -0.6 (1.18)
  Week 36, OC; n=73 | -0.7 (1.13)
  Week 40, LOCF; n=92 | -0.5 (1.24)
  Week 40, OC; n=70 | -0.6 (1.22)
  Week 44, LOCF; n=92 | -0.5 (1.16)
  Week 44, OC; n=69 | -0.6 (1.11)
  Week 48, LOCF; n=92 | -0.6 (1.19)
  Week 48, OC; n=69 | -0.7 (1.14)
  Week 52/EW, LOCF; n=92 | -0.8 (1.19)
  Week 52/EW, OC; n=87 | -0.8 (1.19)

16. Secondary Outcome: Hamilton Rating Scale for Depression (HAM-D) Scale Total Score at Weeks 6, 16, 28, 40, and 52/EW
Description: The HAMD-17 is a 17-item questionnaire that detects change and measures illness severity. Individual items were rated on a scale of 0-4 and 0-2, with the total HAMD-17 score ranging from 0 (not ill) to 52 (severely ill).
Time Frame: Weeks 6, 16, 28, 40, and 52/EW
Population: as for outcome 15
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Lamotrigine
Number analyzed (Participants) | 91
scores on a scale
  Week 6, LOCF; n=91 | 5.2 (6.68)
  Week 6, OC; n=84 | 4.3 (4.85)
  Week 16, LOCF; n=91 | 6.1 (7.28)
  Week 16, OC; n=78 | 5.2 (6.01)
  Week 28, LOCF; n=91 | 5.5 (6.76)
  Week 28, OC; n=77 | 4.5 (5.13)
  Week 40, LOCF; n=91 | 5.9 (7.21)
  Week 40, OC; n=70 | 4.7 (5.53)
  Week 52/EW, LOCF; n=91 | 5.5 (7.30)
  Week 52/EW, OC; n=87 | 5.4 (7.38)

17. Secondary Outcome: Change From Baseline in the Hamilton Rating Scale for Depression (HAM-D) Scale Total Score at Weeks 6, 16, 28, 40, and 52/EW
Description: The HAMD-17 is a 17-item questionnaire that detects change and measures illness severity. Individual items were rated on a scale of 0-4 and 0-2, with the total HAMD-17 score ranging from 0 (not ill) to 52 (severely ill). Change from baseline was calculated as the values at Week 6, 16, 28, 40, and 52 (or EW) minus the baseline value (Week 0).
Time Frame: Baseline (Week 0) and Weeks 6, 16, 28, 40, and 52/EW
Population: as for outcome 15
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Lamotrigine
Number analyzed (Participants) | 91
scores on a scale
  Week 6, LOCF; n=91 | -4.5 (7.37)
  Week 6, OC; n=84 | -4.7 (7.19)
  Week 16, LOCF; n=91 | -3.7 (7.51)
  Week 16, OC; n=78 | -3.8 (7.51)
  Week 28, LOCF; n=91 | -4.3 (7.62)
  Week 28, OC; n=77 | -4.5 (7.66)
  Week 40, LOCF; n=91 | -3.9 (7.77)
  Week 40, OC; n=70 | -3.9 (7.69)
  Week 52/EW, LOCF; n=91 | -4.3 (7.17)
  Week 52/EW, OC; n=87 | -4.1 (6.96)

18. Secondary Outcome: Young Mania Rating Scale (YMRS) Total Score at Weeks 6, 16, 28, 40, and 52/EW
Description: The YMRS is an 11-item, multiple-choice diagnostic questionnaire used to measure the severity of disease in participants. Individual items (1=elevated mood, 2=increased motor activity, 3=sexual interest, 4=sleep, 5=irritability, 6=speech, 7=language thought disorder, 8=content, 9=disruptive aggressive behaviour, 10=appearance, 11=insight) were rated on a scale of 0-4 and 0-8. For all items, 0 is the "best" rating and 4 or 8 is the "worst" rating. YMRS total score was computed as the sum of the scores for the 11 items on the scale. The possible total scores range from 0 (best) to 60 (worst).
Time Frame: Weeks 6, 16, 28, 40, and 52/EW
Population: as for outcome 15
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Lamotrigine
Number analyzed (Participants) | 91
scores on a scale
  Week 6, LOCF; n=91 | 3.2 (6.20)
  Week 6, OC; n=84 | 2.6 (4.37)
  Week 16, LOCF; n=91 | 2.6 (5.83)
  Week 16, OC; n=78 | 1.7 (3.02)
  Week 28, LOCF; n=91 | 2.8 (6.96)
  Week 28, OC; n=77 | 2.0 (5.19)
  Week 40, LOCF; n=91 | 2.7 (6.24)
  Week 40, OC; n=70 | 1.7 (3.95)
  Week 52/EW, LOCF; n=91 | 1.9 (5.55)
  Week 52/EW, OC; n=87 | 2.0 (5.66)

19. Secondary Outcome: Change From Baseline in the Young Mania Rating Scale (YMRS) Total Score at Weeks 6, 16, 28, 40, and 52/EW
Description: The YMRS is an 11-item, multiple-choice diagnostic questionnaire used to measure the severity of disease in participants. Individual items (1=elevated mood, 2=increased motor activity, 3=sexual interest, 4=sleep, 5=irritability, 6=speech, 7=language thought disorder, 8=content, 9=disruptive aggressive behaviour, 10=appearance, 11=insight) were rated on a scale of 0-4 and 0-8. YMRS total score (range of 0-60) was computed as sum of the scores for the 11 items on the scale. Change from baseline was calculated as the values at Week 6, 16, 28, 40, and 52 (or EW) minus the baseline value (Week 0).
Time Frame: Baseline (Week 0) and Weeks 6, 16, 28, 40, and 52/EW
Population: as for outcome 15
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Lamotrigine
Number analyzed (Participants) | 91
scores on a scale
  Week 6, LOCF; n=91 | 0.2 (6.64)
  Week 6, OC; n=84 | -0.3 (5.88)
  Week 16, LOCF; n=91 | -0.4 (7.20)
  Week 16, OC; n=78 | -1.3 (6.13)
  Week 28, LOCF; n=91 | -0.2 (6.89)
  Week 28, OC; n=77 | -1.1 (5.75)
  Week 40, LOCF; n=91 | -0.3 (7.56)
  Week 40, OC; n=70 | -1.1 (6.73)
  Week 52/EW, LOCF; n=91 | -1.1 (7.11)
  Week 52/EW, OC; n=87 | -1.1 (7.27)

20. Secondary Outcome: Median Serum Lamotrigine 200 mg Concentration Among Participants With Concomitant Use of Inducer and Without Inhibitor (at the Timing of Blood Sample Collection)
Description: Pharmacokinetic (PK) samples were collected at Weeks 6, 16, 28, 40, 52/EW, and the plasma lamotrigine concentrations were measured. Participants were required to visit the study site without taking the investigational product on the morning of the PK blood sampling. Inhibitors are defined as drugs that inhibit lamotrigine glucuronidation (i.e., valproate). Inducers are defined as drugs that induce lamotrigine glucuronidation (e.g., carbamazepine). The median value presented is the median of all samples collected at Weeks 6, 16, 28, 40, and 52/EW.
Time Frame: from Week 6 to Week 52/EW
Population: Safety Population. Participants who took at least one dose of drugs that induce lamotrigine glucuronidation (e.g., carbamazepine) from the date of the first dose of study medication to the date of the last dose.
Measure: Median (Full Range); unit: Nanograms per milliliter
Arm/Group | Lamotrigine
Number analyzed (Participants) | 1
Nanograms per milliliter | 1605.70 [0.00 to 3238.6]

21. Secondary Outcome: Median Serum Lamotrigine 100 mg and 200 mg Concentration Among Participants With Concomitant Use of Inhibitor (at the Timing of Blood Sample Collection)
Description: PK samples were collected at Weeks 6, 16, 28, 40, 52/EW, and the plasma lamotrigine concentrations were measured. Participants were required to visit the study site without taking the investigational product on the morning of the PK blood sampling. Inhibitors are defined as drugs that inhibit lamotrigine glucuronidation (i.e., valproate). The median value presented is the median of all samples collected at Weeks 6, 16, 28, 40, and 52/EW.
Time Frame: from Week 6 to Week 52/EW
Population: Safety Population. Participants (par.) who took at least one dose of drugs that inhibit lamotrigine glucuronidation (i.e., valproate) from the date of the first dose of study medication to the date of the last dose. A total of 8 par. were analyzed; 1 par. had both 100 and 200 mg data, 4 par. had 100 mg data only, and 3 par. had 200 mg data only.
Measure: Median (Full Range); unit: Nanograms per milliliter
Arm/Group | Lamotrigine
Number analyzed (Participants) | 8
Nanograms per milliliter
  Lamotrigine 100 mg; n=5 | 5312.30 [3762.7 to 15107.0]
  Lamotrigine 200 mg; n=4 | 6935.40 [3210.2 to 9300.9]

22. Secondary Outcome: Median Serum Lamotrigine 25, 100, 125, 150, 200, 225, 300, and 400 mg Concentrations Among Participants Without Concomitant Use of Inhibitor and Inducer
Description: PK samples were collected at Weeks 6, 16, 28, 40, 52/EW, and the plasma lamotrigine concentrations were measured. Participants were required to visit the study site without taking the investigational product on the morning of the PK blood sampling. Inhibitors are defined as drugs that inhibit lamotrigine glucuronidation (i.e., valproate). Inducers are defined as drugs that induce lamotrigine glucuronidation (e.g., carbamazepine). The median value presented is the median of all samples collected at Weeks 6, 16, 28, 40, and 52/EW.
Time Frame: from Week 6 to Week 52/EW
Population: Safety Population. Participants without concomitant use of inhibitor and inducer from the date of the first dose of study medication to the date of the last dose. Multiple blood samplings were conducted for some participants. A total of 82 participants were analyzed; 4 participants did not have 200 mg dose data but had data for lower doses.
Measure: Median (Full Range); unit: Nanograms per milliliter
Arm/Group | Lamotrigine
Number analyzed (Participants) | 82
Nanograms per milliliter
  Lamotrigine 25 mg; n=2 | 699.95 [527.8 to 872.1]
  Lamotrigine 100 mg; n=12 | 2793.55 [1486.7 to 7440.8]
  Lamotrigine 125 mg; n=1 | 3505.30 [3505.3 to 3505.3]
  Lamotrigine 150 mg; n=1 | 5418.40 [5418.4 to 5418.4]
  Lamotrigine 200 mg; n=78 | 4092.30 [131.0 to 11053.2]
  Lamotrigine 225 mg; n=1 | 3594.25 [2879.3 to 4309.2]
  Lamotrigine 300 mg; n=7 | 5127.10 [3349.4 to 12066.6]
  Lamotrigine 400 mg; n=4 | 8600.40 [4722.2 to 10830.3]

ADVERSE EVENTS:
Arm/Group | Lamotrigine
Serious Adverse Events (participants affected / at risk) | 13/92
Other Adverse Events (participants affected / at risk) | 52/92
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Lamotrigine (N=92)
Gastric cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Mania (Psychiatric disorders) | 4
Depression (Psychiatric disorders) | 2
Delirium (Psychiatric disorders) | 1
Self injurious behaviour (Psychiatric disorders) | 1
Suicidal ideation (Psychiatric disorders) | 1
Sick sinus syndrome (Cardiac disorders) | 1
Pharyngitis (Infections and infestations) | 1
Abortion spontaneous (Pregnancy, puerperium and perinatal conditions) | 1
Ovarian hemorrhage (Reproductive system and breast disorders) | 1
Asthma (Respiratory, thoracic and mediastinal disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Lamotrigine (N=92)
Nasopharyngitis (Infections and infestations) | 36
Abdominal pain upper (Gastrointestinal disorders) | 14
Stomatitis (Gastrointestinal disorders) | 11
Nausea (Gastrointestinal disorders) | 7
Vomiting (Gastrointestinal disorders) | 7
Diarrhea (Gastrointestinal disorders) | 6
Headache (Nervous system disorders) | 6
Anemia (Blood and lymphatic system disorders) | 5
Back pain (Musculoskeletal and connective tissue disorders) | 5

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.